CLINICAL TRIAL: NCT05212714
Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) to Reduce Post Traumatic Stress Disorder (PTSD) Symptoms in World Trade Center (WTC) Responders
Brief Title: taVNS to Reduce PTSD Symptoms in WTC Responders
Acronym: taVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Rebecca Schwartz, Associate Professor and Chief, Social Behavioral Sciences, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 21-0640; U01OH012050 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2022-01-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: feasibility and acceptability; WTC responders; taVNS
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study seeks to conduct a randomized, double-blind placebo-controlled parallel-design pilot study, to determine whether the taVNS intervention and study methodology are feasible and acceptable for use with WTC responders with PTSD. It is important that the design is double-blind and placebo-controlled in order to have the most appropriate control and to limit bias on the part of the participant and investigators. In addition, as this is a feasibility study, it is important to replicate the methodology that will eventually be used with a larger trial in order to truly assess whether the intervention and methodology are acceptable, feasible and efficacious.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- taVNS Treatment (Experimental): n = 20
  Interventions: Device: taVNS
- Sham Comparator (Sham Comparator): n = 10
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — The non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) device that will be used in this study is a wearable TENS unit called the Vorso STIM100 System. The Vorso system consists of a wearable, external stimulator, a neural interface ear piece, and an arm band designed to be safe for human contact. The external stimulator generates electrical pulses that are transcutaneously delivered to the auricular branch of the vagus nerve through the ear canal. The ear piece contains 4 electrodes that carry current from the external stimulator to the auricular branch of vagus nerve. The external stimulator connects to a flexible arm band that attaches to the upper arm for ease of use during each stimulation session. The type of stimulation (including shape, frequency, pulse width, amplitude, total charge, and energy delivered) is comparable to the levels applied by commercially available TENS stimulators. The sham control group will not receive any stimulation.

SUMMARY:
This study seeks to conduct a randomized, double-blind pilot study, to determine whether the Transcutaneous Auricular Vagus Nerve Stimulation and study procedure are feasible and acceptable for use with World Trade Center responders with Post Traumatic Stress Disorder.

DETAILED DESCRIPTION:
Participants will be randomized to one of two groups; one that receives stimulation and one that does not. Once their device is ready (roughly 1 month), they will be asked to participate in a baseline questionnaire. They will also be given a phone to interface with the device and record their usage and will use the device for one 15-minute session under the supervision of members of the research team and be monitored using a combination of non-invasive equipment, including an brain activity monitoring cap, blood pressure cuff (to monitor blood pressure), a respiratory belt (to monitor respirations) and an eye tracking device (to monitor eye movement). Researchers are using these tests to see if there are any inflammatory, neural, and cardiovascular changes that relate to the treatment. A research nurse will collect 12 mL of blood (roughly 2 tsp) before and after their session. Blood will be drawn to look at markers of inflammation before using the device, after using the device, and again at the 6-week follow-up visit. They will then be asked to complete a survey regarding the stimulation device on an iPad. After their initial visit, they will be instructed to use the device twice a day, every day at home, for 15 minutes over 8 weeks. After 8 weeks, they will be asked to come in for a final visit, where they will be asked to complete another 15-minute device session, blood draw and survey regarding their experiences.

ELIGIBILITY:
Inclusion Criteria:

* being a Queens WTCHP responder who agreed to be contacted to participate in research
* having PTSD as per DSM criteria indicated by the GRDC
* having elevated PTSD symptoms, indicated by a PCL-S93 score > 44 during an annual monitoring visit between 2018-2020
* having a score of 33 or greater on the PCL-594 delivered during the initial phone screen to determine current symptomatology
* meeting diagnostic indication of PTSD using a Clinician-Administered PTSD Scale (CAPS), which is a clinical interview assessment.95

Exclusion criteria:

* being physically/mentally unable to consent and participate
* inability to speak, read, or write in English,
* exhibiting any current psychotic or manic symptoms, active substance dependence, or current suicidal or homicidal intent/plan, as per the standard MINI neuropsychological assessment.96
* active disease involving the auricle or ear canal (e.g., otitis media, tinnitus, infection, perforated tympanic membrane, vestibular and/or balance, excessive cerumen production, skin irritation), unwilling to remove a piercing (e.g., daith or tragus), or use a device (e.g., hearing aid, cochlear implant) that would preclude daily use of the earpiece.
* history of unilateral or bilateral vagotomy.
* Current pregnancy (self-report)
* previously implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators, VNS).
* other major conditions, that in the judgment of the investigators/WTCHP medical staff, would make the participant unsuitable for inclusion or would interfere with the participant participating in or completing the study. these include:

  * current treatment with psychotropic medication, including tricyclics, antipsychotics, mood stabilizers, bupropion, barbiturates, stimulants, antiepileptics, opioid medications.
  * current diagnosis or history of any clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, neurologic, gastrointestinal, or immunologic.
  * history of any of the following cardiovascular conditions: Moderate to severe congestive heart failure (New York Heart Association class III or IV); Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting; Uncontrolled hypertension as defined by a confirmed systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
  * history of or active seizure disorder.
  * history of recurrent vasovagal syncope episodes.
  * diagnosis of cancer (other than non-invasive skin cancer or carcinoma in-situ of the cervix) within the 5 years prior to study entry.
  * history of concurrent illness that requires hospitalization within 30 days prior to study entry
  * have hypertension/hypotension uncontrolled by medication
  * participation in another investigational trial during the 30 days prior to study entry or during this project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of Utilizing taVNS with WTCHP Responders as Measured By Rates of Recruitment | 8 week follow-up
  Evaluated as: (1) rates of recruitment (per month)
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.
Feasibility of Utilizing taVNS with WTCHP Responders as Measured By Intervention Adherence | 8 week follow-up
  Evaluated as: (2) adherence to the taVNS intervention
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.
Feasibility of Utilizing taVNS with WTCHP Responders as Measured By Retention Rates | 8 week follow-up
  Evaluated as: (3) 8-week retention
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.
Feasibility of Utilizing taVNS with WTCHP Responders as Measured By Duration | 8 week follow-up
  Evaluated as: (4) duration of study assessments
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.
Feasibility of Utilizing taVNS with WTCHP Responders as Measured By Completion Rates | 8 week follow-up
  Evaluated as: (5) completion rate of study assessments
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.

SECONDARY OUTCOMES:
Acceptability of taVNS by WTCHP Responders As Assessed by Time to Completion of Questionnaires and Biological Data | 8 week follow-up
  Assessing: (1) the time to completion of questionnaires and biological data/blood draw
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.
Acceptability of taVNS by WTCHP Responders As Assessed by Percentage Missing Data | 8 week follow-up
  Assessing: (2) percentage of missing data from questionnaires
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.
Acceptability of taVNS by WTCHP Responders As Assessed by Rate of Refusal | 8 week follow-up
  Assessing: (3) the rate of refusal of biologic measurements and blood draw
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.
Acceptability of taVNS by WTCHP Responders As Assessed by Score of taVNS Satisfaction and Usefulness Questionnaire | 8 week follow-up
  Assessing: (4) the score on the taVNS Satisfaction and Usefulness Questionnaire
  All measures will be described using frequency and percent or mean (SD) as appropriate, overall and by taVNS and sham group, with corresponding 95% confidence intervals to interpret the precision of the estimates. Median and interquartile range may also be used if discrete data are skewed.

OTHER OUTCOMES:
Mental Health Measures | Baseline and 8 week follow-up
  Tertiary outcome measures validated self-report mental health measures.
  For all tertiary outcomes, descriptive statistics for each time point, as well as differences over time, will be calculated. Differences in outcomes will be assessed from the first time point at baseline and the last time point at 8 weeks, for long-term effects. Within-subject correlation of acute and long-term measures will be reported.
PTSD | Baseline and 8 week follow-up
  Tertiary outcome measures include the administration of the CAPS PTSD interview.
  For all tertiary outcomes, descriptive statistics for each time point, as well as differences over time, will be calculated. Differences in outcomes will be assessed from the first time point at baseline and the last time point at 8 weeks, for long-term effects. Within-subject correlation of acute and long-term measures will be reported.
Biologic Potential Endpoints - Heart Rate | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures such as heart rate.
  • Heart rate/HRV (6-lead ECG, DI Powerlab) (beats/min, range=40-150)
  The 6-lead electrocardiogram (ECG) will be recorded from wires connected from a bio-amplifier to four foam electrodes that are adhesively attached to the left shoulder, the right shoulder, the left ankle, and the right ankle. The right ankle provides a ground, while the remaining three leads provide recordings of the electrical potentials between different sites that represent the electrical activity of the heart in real-time.
  The vitals will be collected by the ADInstruments PowerLab, ADInstrument sensors for collecting human physiological signals, and corresponding Labchart software.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Biologic Potential Endpoints - Galvanic Skin Response | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures such as galvanic skin response.
  • Galvanic Skin Response (GSR electrodes, ADI Powerlab) (skin conductance in microSiemens, range=0-50mS)
  The vitals will be collected by the ADInstruments PowerLab, ADInstrument sensors for collecting human physiological signals, and corresponding Labchart software.
  Two additional sensors are placed on the left wrist and hand of the participant. The first set records electrodermal activity (EDA) by attaching two dry, metal electrodes with Velcro attachments on two fingers, preferably the pointer and ring fingers on the dominant hand. These electrodes measure the changes in skin conductance that can reflect changes in sweat gland activity.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Biologic Potential Endpoints - Skin Temperature | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures such skin temperature.
  • Skin Temperature (Thermistor Pod, ADI Powerlab) (Celsius, range=30-35C)
  The vitals will be collected by the ADInstruments PowerLab, ADInstrument sensors for collecting human physiological signals, and corresponding Labchart software.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Biologic Potential Endpoints - Respiratory Rate | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures such respiratory rate.
  • Respiratory Rate (Respiratory Belt, ADI Powerlab) (breaths per minute, range=3-20BPM)
  The vitals will be collected by the ADInstruments PowerLab, ADInstrument sensors for collecting human physiological signals, and corresponding Labchart software.
  A respiratory belt that goes around the torso will be attached to the participant and is tightened without discomfort such that breathing causes the belt to stretch, which provides inspiration (inhalation) and expiration (exhalation) times to infer respiration rate.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Biologic Potential Endpoints - Blood Pressure | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures such as beat-to-beat blood pressure.
  • Beat-to-Beat Blood Pressure (Human Non-Invasive Blood Pressure Nano Interface, ADI Powerlab) (mmHg, range=50-150mmHg)
  A wrist device will be placed to record non-invasive blood pressure (NIBP) from the participant's left hand. The wrist device is placed with a Velcro strap on the wrist, while a small cuff is placed on the middle finger. The wrist device provides air and power for the cuff to inflate and deflate to measure changes in blood pressure.
  The vitals will be collected by the ADInstruments PowerLab, ADInstrument sensors for collecting human physiological signals, and corresponding Labchart software.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Biologic Potential Endpoints - EMG | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures such as EMG.
  • Facial & Neck Electromyography (EMG electrodes, ADI Powerlab) (millivolts, range=0-15mV)
  Electromyogram (EMG) will be recorded by placing foam adhesive electrodes on the participant's neck. Leads are connected from these electrodes to the same bio-amplifier as the ECG.
  The vitals will be collected by the ADInstruments PowerLab, ADInstrument sensors for collecting human physiological signals, and corresponding Labchart software.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Biologic Potential Endpoints - EEG | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures of EEG(DSI-24) (band-power dB changes, range=0-10)
  Electroencephalography will be collected by a DSI-24 cap developed by Wearable Sensing, which offers low noise and high signal quality of non-invasive brain recordings.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Biologic Potential Endpoints - Pupil Dilation | Baseline and 8 week follow-up
  Tertiary outcome measures include biological measures of pupil dilation (Tobii Pro Glasses 2) (pupil diameter in mm, range=2-8mm).
  The eye tracking glasses, the Tobii Pro Glasses 2 are easily wearable and mobile glasses with multiple small cameras to track gaze location and pupil size.
  All biological measures will be administered at the baseline visit 10 minutes before using the device and after using the device at the 8 week follow-up visit. All data will be compiled and analyzed using MATLAB.
Markers of Inflammation - TNFα, (IL)-1β, IL-6, IL-10, IL-12, IL-17, CRP, cortisol, and alpha amylase | Baseline and 8 week follow-up
  Tertiary outcome measures a blood draw to assess markers of inflammation before using the device at baseline and after using the device at the 8 week follow-up visit. Inflammatory markers include Tumour Necrosis Factor alpha (TNFα), Interleukin (IL)-1β, IL-6, IL-10, IL-12, IL-17, C Reactive Protein (CRP), cortisol, and alpha amylase.
  For all tertiary outcomes, descriptive statistics for each time point, as well as differences over time, will be calculated. Differences in outcomes will be assessed from the first time point at baseline and the last time point at 8 weeks, for long-term effects. Within-subject correlation of acute and long-term measures will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schwartz, PhD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institutes for Medical Research, Manhasset, New York, United States

DOCUMENTS (1):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT05212714/Prot_000.pdf